CLINICAL TRIAL: NCT03434444
Title: In Vitro Optimization of Oxytocin-induced Myometrial Contractility by Propranolol - Potential Applications in Induction of Labour and Treatment of Postpartum Hemorrhage
Brief Title: In Vitro Optimization of Oxytocin-induced Myometrial Contractility by Propranolol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-04
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Postpartum Hemorrhage
Keywords: propranolol; oxytocin; uterine contraction
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Low Dose Oxytocin (Active Comparator): The myometrial samples are bathed in an oxytocin solution at increasing concentrations (from 10 -12M to 10 -9M)
  Interventions: Drug: Oxytocin
- Propranolol (Active Comparator): The myometrial samples are bathed in a propranol solution at 10 -6M
  Interventions: Drug: Propranolol
- Propranolol + low dose oxytocin (Active Comparator): The myometrial samples are bathed in an oxytocin solution at increasing concentrations (from 10 -12M to 10 -9M) plus propranol (10 -6M)
  Interventions: Drug: Oxytocin; Drug: Propranolol
- High Dose Oxytocin (Active Comparator): The myometrial samples are bathed in an oxytocin solution (10 -5M), followed by increasing concentrations of oxytocin (from 10 -8M to 10 -5M)
  Interventions: Drug: Oxytocin
- High Dose Oxytocin, Propranolol-pretreated (Active Comparator): The myometrial samples are bathed in an oxytocin solution (10 -5M) plus propranolol (10 -6M), followed by increasing concentrations of oxytocin (from 10 -8M to 10 -5M)
  Interventions: Drug: Oxytocin; Drug: Propranolol
- High dose oxytocin + propranolol (Active Comparator): The myometrial samples are bathed in an oxytocin solution (10 -5M), followed by increasing concentrations of oxytocin (from 10 -8M to 10 -5M) plus propranolol (10 -6M)
  Interventions: Drug: Oxytocin; Drug: Propranolol

INTERVENTIONS:
Drug: Oxytocin — Oxytocin in solution, ranging from 10 -12M to 10 -5M
  Other Names: pitocin
  Arms: High Dose Oxytocin; High Dose Oxytocin, Propranolol-pretreated; High dose oxytocin + propranolol; Low Dose Oxytocin; Propranolol + low dose oxytocin
Drug: Propranolol — Propranolol in solution, 10-6M
  Arms: High Dose Oxytocin, Propranolol-pretreated; High dose oxytocin + propranolol; Propranolol; Propranolol + low dose oxytocin

SUMMARY:
The rates of cesarean deliveries (CD) and postpartum hemorrhage (PPH) are on the rise, with failed induction and augmentation of labor as major contributing factors. Oxytocin is commonly used for labor induction, as well as during the third stage of labor to minimize the risk of primary PPH. At delivery, it is imperative that the uterus responds effectively to parenteral oxytocin. Poor response to oxytocin following delivery is commonly due to prolonged labor with oxytocin augmentation that is known to "desensitize" the myometrium. Despite the option of several second line uterotonic agents, none of them are as effective as oxytocin in controlling PPH. Given that poor uterine muscle contraction is the root cause of both failed induction or augmentation (leading to a CD in labor) and uterine atony (leading to PPH), there is an urgent and clinically important need to investigate novel methods to enhance oxytocin-induced myometrial contractions.

Propranolol, a beta adrenergic receptor agonist, has the potential to improve myometrial contractions by virtue of its ability to inhibit catecholamine production. The investigators plan to investigate the effects of propranolol in both naive and desensitized myometrium, in order to better understand its potential role in improving labor induction and reducing the risk of PPH following oxytocin exposure during labor.

The investigators hypothesize that propranolol is likely to potentiate the action of oxytocin upon human myometrium, to ultimately help improve the success of labor induction/augmentation and treatment of PPH.

DETAILED DESCRIPTION:
Myometrial samples will be used to investigate the effect of propranolol on uterine contractions when exposed to high and low doses of oxytocin (to simulate PPH treatment and labor induction respectively).

The tissue will also be frozen at the end of the experiment, and Western blotting will be used to investigate the effect of propranolol on the expression patterns and cellular distribution of the oxytocin receptor and beta-adrenergic receptor and their signaling pathways in desensitized myometrium.

ELIGIBILITY:
Inclusion Criteria:

* Patients who give written consent to participate in this study
* Patients with gestational age 37-41 weeks
* Non-laboring patients, not exposed to exogenous oxytocin
* Patients requiring primary Cesarean delivery or first repeat Cesarean delivery

Exclusion Criteria:

* Patients who refuse to give written informed consent
* Patients who require general anesthesia
* Patients who had previous uterine surgery or more than one previous Cesarean delivery
* Patients with any condition predisposing to uterine atony and postpartum hemorrhage, such as abnormal placentation, multiple gestation, preeclampsia, macrosomia, polyhydramnios, uterine fibroids, bleeding diathesis, chorioamnionitis, or a previous history of postpartum bleeding
* Emergency Cesarean section in labor
* Patients on medications that could affect myometrial contractility, such as nifedipine, labetolol or magnesium sulfate

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Motility index | 3 hours
  Motility index (MI) takes into account both the amplitude and frequency of the myometrial contraction. It is a calculated outcome, based on the formula: frequency/(10 x amplitude).
  The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.

SECONDARY OUTCOMES:
Amplitude of contraction | 3 hours
  The maximum extent of uterine muscle contraction, measured in grams (g). The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Frequency of contraction | 3 hours
  The number of contractions in uterine muscle (myometrium) over 10 minutes, spontaneously and in response to an agonist.
  The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Integrated area under response curve (AUC) | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Balki M, Miller LM, Caliaperumal J, Wang S, Huszti E, Kingdom JC. Propranolol and Oxytocin-Induced Contractility in Gravid Human Myometrium: An Ex Vivo Laboratory Study. BJOG. 2025 Aug;132(9):1228-1237. doi: 10.1111/1471-0528.18146. Epub 2025 Mar 24. PMID 40129234